

| Official Title: | Evaluating Smoking Cessation and Harm Reduction Approaches Among People Living With HIV/AIDS in South Africa |
|---|---|
| NCT Number: | NCT06169813 |
| Study Number: | 22-00868 |
| Document Type: | Informed Consent Form |
| Date of the Document: | • April 4, 2023 |



PLACE BARCODE STICKER

## In accordance with the provisions of the Protection of Personal Information Act 4 of 2013 (as amended), I hereby consent:

- a. To my personal information (hereinafter 'data') being collected, processed, shared and stored in accordance with the research protocol as approved by the South African Medical Research Council's Human Research Ethics Committee (SAMRC HREC);
- b. To my anonymised data being shared, processed and transferred by third parties and between third parties, and where relevant beyond the jurisdictional borders of South Africa;
- c. To all findings and results flowing from my anonymised data being broadly shared and published on the conclusion of the research.

## I am aware of the risks of the study, which are as follows:

Risks of Nicotine Replacement Therapy:

Using nicotine replacement therapy may result in the following:

- some stomach discomfort or dizziness,
- headaches,
- insomnia (trouble falling or staying asleep),
- rapid heartbeat,
- or skin irritation when using patches

## Risks of E-Cigarettes:

The use of e-cigarettes has shown an increased risk of health problems if used consistently in conjunction with cigarettes. You should aim to totally switch to e-cigarettes by the end of the intervention and you should NOT use other brands of e-cigarettes while you are participating in this study. Use of E-Cigarettes may cause the following:

- nausea or vomiting,
- abdominal pain,
- throat or eye irritation,
- insomnia,
- dizziness

## I declare that:

- I have read or had read to me this information and consent form and it is written in a language with which I am fluent and comfortable.
- I am older than 18 years of age
- I have had a chance to ask questions and all my questions have been adequately answered.
- I know that taking part in this study is voluntary and I have not been forced to take part. I may choose to leave the study at any time without any problems.

| Signed at: | on (date) |
|---|---|
| Name of participant | Signature of participant |
| Name of witness | Signature of witness |
| Declaration by investigato | |
| | declare that I have explained the i |
| | I have encouraged him/her to ask qu<br>hem. I am satisfied that he/she adequately understands<br>ve. |
| Signed at: | on (date) |
| Name of investigator | Signature of investigator |